CLINICAL TRIAL: NCT03732183
Title: A Brief Mind-Body Program to Support Military and Veteran Caregiver Wellness: a Pilot Study
Brief Title: A Podcast Mind-Body Program for Military Caregiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Elizabeth Dole Foundation (Unknown)
Responsible Party: Principal Investigator, Eric Bui, MD, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017P002426
Record Dates: First submitted 2018-06-26; First posted 2018-11-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Stress, Psychological
Keywords: Stress; Military Caregiver; Caregiver; Online; Podcast; Mind-Body; Wellness
MeSH Terms: conditions — Stress, Psychological | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Podcast SMART-3RP (Experimental): The mind body intervention is delivered by podcast and material posted online. All session content will be audio recorded into 15-min audio-recordings that will be delivered on a podcast platform. During the course of the 4-week program, one new "podcast session" will be delivered every day.
  Interventions: Behavioral: Podcast SMART-3RP

INTERVENTIONS:
Behavioral: Podcast SMART-3RP — 28 daily podcasts, each 15 minutes.
  Other Names: SMART-3RP; Meditation

SUMMARY:
The purpose of this pilot study is to test the efficacy, feasibility, and acceptability of a brief, online, mind-body wellness program to reduce stress and promote resilience in military caregivers.

DETAILED DESCRIPTION:
The investigators are piloting a brief, online, mind-body program to reduce stress in military caregivers. Eligible participants are, 1) At least 18 years old 2) Serving as military caregivers and 3) have regular access to a smartphone or computer. The investigators have adapted the SMART-3RP into a brief podcast, which we plan to administer daily. Participants will be administered questionnaires at baseline, mid-program, and post-program to assess for symptoms of stress, anxiety, and depression. Participants will be compensated for completing all measures.

ELIGIBILITY:
Inclusion Criteria:

* Military Caregivers
* 18 years of age
* Regular Access to smartphone or computer

Exclusion Criteria:

* Non-Military Caregivers
* Under 18 years of age
* No regular access to smartphone or computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | 1 month
  total score ranges 0-40

SECONDARY OUTCOMES:
Patient Health Questionnaire-8 (PHQ-8) | 1 month
  score ranges from 0-24
Generalized Anxeity Disorder-7 (GAD-7) | 1 month
  score ranges from 0-21
Medical Symptom Checklist (MSCL) | 1 month
  score ranges from 0-175
PROMIS - Satisfaction with Participation in Social Roles - Short Form (SPSR): | 1 month
  raw scores range from 8-40
PROMIS - Ability to Participate in Social Roles and Activities - Short Form 4A (ASPRA): | 1 month
  raw scores range from 4-20

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bui, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MassGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No